CLINICAL TRIAL: NCT02330302
Title: A Randomized Controlled Trial Comparing Single Shot Fascia Iliaca Block With Femoral Nerve Block for Analgesia Following Surgical Fixation of Hip Fractures
Brief Title: Single Shot Fascia Iliaca Block vs Femoral Nerve Block for Analgesia for Surgical Fixation of Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/453/D
Record Dates: First submitted 2014-12-31; First posted 2015-01-01 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral nerve block (Active Comparator): Procedure: Ultrasound-guided femoral nerve block Drug: Ropivacaine 0.5% 30mls
  Interventions: Drug: Ropivacaine
- Fascia Iliaca block (Active Comparator): Procedure: Ultrasound-guided suprainguinal approach to fascia iliaca block Drug: Ropivacaine 0.5% 30mls
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Ultrasound-guided femoral nerve block with Ropivacaine 0.5% 30mls
  Other Names: naropin
  Arms: Femoral nerve block
Drug: Ropivacaine — Ultrasound-guided suprainguinal approach to fascia iliaca block with Ropivacaine 0.5% 30mls
  Other Names: naropin
  Arms: Fascia Iliaca block

SUMMARY:
Hip fractures are common in our elderly population and is associated with pain before and after surgery. The current pain management for patients who have undergone surgery for hip fractures include a combination of oral painkillers, opioids (eg morphine) and regional anaesthesia techniques, which involves the injection of local anaesthetic drugs near nerves supplying the hip joint to numb the operation site. As opioids have many side effects, especially in the elderly patients, regional anaesthesia techniques can help to reduce the use of opioids and the related side effects. This may enhance their recovery and length of hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgical fixation of hip fracture
* Patients with isolated inter-trochantric fracture
* American Society of Anesthesiologists (ASA) physical status 1 to 3
* Patients who are able to give their own consent

Exclusion Criteria:

* Patients unable to give consent or inability to communicate/ cooperate
* Patients with regular consumption of strong opioids (morphine, oxycodone) or steroids
* Patients with allergy to local anaesthetics or any drugs included in the study
* Patients with contraindications to spinal anaesthesia such as coagulation disorders/ thrombocytopenia and local infection at site of injection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain scores | up to 24 hours
  resting and dynamic pain scores are obtained pre-intervention, 30mins post intervention (and on positioning for spinal anaesthesia), 1 hr post-operatively and at 24hrs post intervention

SECONDARY OUTCOMES:
opioid requirement/consumption | for first 24 hrs (including intra operatively) following intervention
  need for additional opioids during first 24hrs following intervention record of any opioid related side effects will be kept as well

OTHER OUTCOMES:
complications associated with intervention | at 24 hrs post intervention
  including hematoma, infection, prolonged neurologic deficits, occurence of falls

CONTACTS AND LOCATIONS:
Overall Officials: Yean Chin Lim, MBBS, MMed, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore